CLINICAL TRIAL: NCT00756197
Title: A Single Center Pilot Study of CryoSpray Ablation(TM) to Determine Safety and Feasibility in Radiation Induced Proctitis (CSA LGI-2)
Brief Title: CryoSpray Ablation(TM)to Determine Safety and Feasibility in Radiation Induced Proctitis
Acronym: CSALGI2
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Considering more robust design.
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00016-00
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Radiation Proctitis; Radiation Induced Proctitis
Keywords: Radiation Proctitis; Radiation Induced Proctitis
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryo Spray Ablation Group 1 (Experimental): 4 cycles of 10 seconds each
  Interventions: Device: Cryo Spray Ablation Group 1
- Cryo Spray Ablation Group 2 (Experimental): 2 cycles of 20 seconds each
  Interventions: Device: Cryo Spray Ablation Group 2

INTERVENTIONS:
Device: Cryo Spray Ablation Group 1 — Cryo Spray Ablation
  Other Names: CryoSpray Ablation; Cryospray; Cryotherapy; Cryo Spray Ablation
  Arms: Cryo Spray Ablation Group 1
Device: Cryo Spray Ablation Group 2 — cryo spray ablation
  Arms: Cryo Spray Ablation Group 2

SUMMARY:
The purpose of this study is to evaluate the safety, feasibility, tissue response, and subject side effects of liquid nitrogen sprayed through a catheter (CryoSpray AblationTM, "CSA" or "cryospray therapy") via endoscope in subjects with radiation induced proctitis.

DETAILED DESCRIPTION:
The proposed study is a single center, ten patient pilot study to evaluate the safety and feasibility of sprayed liquid nitrogen through a catheter via endoscope in subjects with radiation proctitis. There will be two groups. Subjects in Group 1 will receive a cryospray applied to healthy tissue for 10 seconds. The cryospray will be repeated four (4) times in sequential fashion for a total of 40 seconds of cryospray therapy. Subjects in Group 2 will receive a cryospray applied to healthy tissue for 20 seconds. The cryospray will be repeated two (2) times in sequential fashion for a total of 40 seconds of cryospray therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age
* Have radiation induced proctitis

Exclusion Criteria:

* Pregnant or nursing
* Planning to become pregnant during the course of the study
* Planning to sire a child while enrolled in the study
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.

Subject has prior or concurrent ablation therapy including, but not limited to, photodynamic therapy, multipolar electro coagulation, argon plasma coagulation, laser treatment, radio frequency, etc

* Refusal or inability to give consent.
* Concurrent chemotherapy.
* Medical contraindication or potential problem that would preclude study participation
* Concurrent participation in other experimental studies
* Uncontrolled coagulopathy or bleeding diathesis
* Portal hypertension due to cirrhosis manifest by esophageal, gastric or rectal varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoints for this study are patient safety, treatment efficacy, and feasibility of cryospray therapy in subjects with radiation proctitis. | End of Study

SECONDARY OUTCOMES:
The secondary endpoints for the study are the cataloging of side effects, and tissue response as determined by endoscopic visual evaluation. | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lee Krinsky, D.O., Principal Investigator — VA San Diego Medical Center

REFERENCES:
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Cash BD, Johnston LR, Johnston MH. Cryospray ablation (CSA) in the palliative treatment of squamous cell carcinoma of the esophagus. World J Surg Oncol. 2007 Mar 16;5:34. doi: 10.1186/1477-7819-5-34. PMID 17367523
- [Background] Pinsonneault C, Fortier J, Donati F. Tracheal resection and reconstruction. Can J Anaesth. 1999 May;46(5 Pt 1):439-55. doi: 10.1007/BF03012943. PMID 10349923
- [Background] Dumot JA. Cryotherapy Ablation for Esophageal HGD or IMCA in High Risk, Non-Surgical Patients. DDW2007 Abstract submission. Cleveland Clinic Foundation (pending publication)
- [Background] Greenwald BD. CryoSpray Ablation of Early Esophageal Cancer. DDW 2007 Abstract submission. University of Maryland Medical Center. (pending publication)
- [Background] Johnston M, Horwhat J, Dubois A, Schoenfeld P. Endoscopic cryotherapy in the swine esophagus: A follow-up study (Abstract). Gastrointestinal Endoscopy 49:AB126, 1999.
- [Background] Johnston MH, Horwhat JD, Haluska, Moses FM. Depth of injury following endoscopic spray cryotherapy: EUS assisted evaluation of mucosal ablation and subsequent healing in the swine model (Abstract). Gastrointestinal Endoscopy 51: AB98, 3462, 2000.
- [Background] Johnston MH. Endoscopic cryotherapy: A new ice age in gastroenterology? Medscape Gastroenterology 2: 187, 2000.
- [Background] Eastone JA, Horwhat D, Haluska O, Mathews J, Johnston M. Cryoablation of swine esophageal mucosa: A direct comparison to argon plasma coagulation (APC) and multipolar electrocoagulation (MPEC) [Abstract] Gastrointestinal Endoscopy 53: A3448, 2001.
- [Background] Johnston MH, Eastone JA, Horwhat JD. Reversal of Barrett's esophagus with cryotherapy [Abstract]. American Journal of Gastroenterology 98(9 Suppl): A30, S11, 2003.
- [Background] Johnston MH, Cash BD, Horwhat JD, Johnston LR, Dykes CA, Mays HS. Cryoablation of Barrett's Esophagus (BE) [Abstract]. Gastroenterology 130 (4, Suppl.2): A640, 2006.
- [Background] Johnston MH, Cash BD, Dykes CA, Mays HS, Johnston LR. Cryoablation of dysplasia in Barrett's Esophagus (BE) and early stage esophageal cancer [Abstract]. Gastrointestinal Endoscopy 63 (5): April, 2006.